CLINICAL TRIAL: NCT02633826
Title: The Role of Pre-formed Alloreactive T Cells on Acute Rejection Episodes and Long-term Graft Outcome in Patients After Living Donor Renal Transplantation
Brief Title: Pre-formed Alloreactivity in Renal Transplant Recipients
Status: Completed | Type: Observational
Sponsor: Martina Sester (Other)
Responsible Party: Sponsor-Investigator, Martina Sester, Univ.-Prof. Dr. Martina Sester, Universität des Saarlandes
Organization: Universität des Saarlandes (Other)
Other Study IDs: Pre-formed alloreactivity
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplantation; Acute Graft Rejection
Keywords: alloreactive T cell; donor-specific antibody

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- kidney transplant recipients: kidney transplant recipients of an allograft from a living donor, no intervention

SUMMARY:
This investigator-initiated study will analyse the role of pre-formed alloreactive T cells on acute rejection episodes and graft outcome in kidney transplant recipients after living donation.

DETAILED DESCRIPTION:
In recipients of solid organ transplants, preformed alloreactive T cells may mediate acute rejections and compromise long-term graft survival. Previous studies on the role of alloreactive T cells in transplantation were hampered by the fact that experimental assays to quantify alloreactivity were technically demanding and not suitable for use in a clinical setting. Based on a recent development of a whole-blood assay, alloreactive T cells may be quantified and characterised within one day. This assay therefore provides the experimental basis to study the development and the role of alloreactive T cells in a clinical setting in patients after renal transplantation. This will be performed in a multicenter study in living donor renal transplant recipients where preformed alloreactivity of the recipient towards the living donor will be determined and associated with standard clinical parameters of graft function and long-term graft outcome on follow-up. In addition, the development of donor-specific antibodies will be analysed after transplantation. If this project was able to provide evidence for a role of alloreactive T cells in acute rejection episodes or long-term graft function, this assay may in future be used to guide individualized immunosuppressive drug treatment early after transplantation. It will thereby aid in distinguishing patients where standard immunosuppressive drug regimens are sufficient from the minor population of patients at high risk for rejection who will benefit from intensified drug regimens.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* First or second renal transplantation
* Living donor renal transplantation
* Recipient older than 18 years
* Negative cross match
* Planed quadruple, Tacrolimus-based (low-dose) immunosuppressive drug regimen (Tacrolimus, 2g MMF starting dose, (methyl)prednisolone according to center practice, basiliximab at day 0 and day 4)
* Planned start of Tacrolimus (Advagraf®) 3 to 10 days prior to transplantation (trough levels 5-10 ng/ml during the first 3 months, 5-7 ng/ml thereafter)

Exclusion Criteria:

* Planed T-cell depleting induction therapy
* Pregnancy
* Pre-existing, moderate to high dose immunosuppressive medication
* Pre-existing, severe lymphopenia (< 400/µl)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Transplant recipients of a kidney from a living donor
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
graft function | 1 year
  1-year graft function (estimated glomerular filtration rate)

SECONDARY OUTCOMES:
Creatinine | 1 year
  1-year creatinine
Cystatin C | 1 year
  1-year cystatin C
rejection: acute rejection episodes within the first year | 1 year
proteinuria within the first year | 1 year

CONTACTS AND LOCATIONS:
Locations (13):
- Germany (13):
  - Saarland University, Homburg, Saarland
  - Medizinische Klinik II, Aachen University, Aachen
  - Charité Berlin, Berlin
  - Klinikum Köln-Lindenthal, Cologne
  - University Erlangen Nürnberg, Erlangen
  - Medizinische Klinik III, Frankfurt University, Frankfurt
  - University Clinic of Giessen and Marburg (UKGM), Giessen
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - Transplantationszentrum Heidelberg - Nephrologie, Heidelberg
  - University of Lübeck, Lübeck
  - University of Mainz, Mainz
  - University of Münster, Münster
  - Innere Medizin IV, University of Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: No